CLINICAL TRIAL: NCT00993824
Title: Use of Continuous Glucose Monitoring With Ambulatory Glucose Profile Analysis to Demonstrate the Glycemic Effect of Colesevelam HCl (Welchol) in Patients With Type 2 Diabetes
Brief Title: Glycemic Effect of Colesevelam HCl (Welchol) in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 03901-09-C
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Welchol then Placebo (Placebo Comparator): 3.75 grams of colesevelam HCl (Welchol) at evening meal for 12 weeks, and then crossover to placebo at evening meal for 12 weeks.
  Interventions: Drug: colesevelam HCl; Drug: placebo
- Placebo then Welchol (Placebo Comparator): Placebo taken for 12 weeks at evening meal, and then crossover to 3.75 grams of colesevelam HCl taken at evening meal fro 12 weeks.
  Interventions: Drug: colesevelam HCl; Drug: placebo

INTERVENTIONS:
Drug: colesevelam HCl — 3.75 grams of colesevelam HCl (6 tablets)
  Other Names: Welchol
Drug: placebo

SUMMARY:
The purpose of this study is to obtain continuous glucose monitoring (CGM) data from individuals taking Welchol compared to placebo. The CGM data will determine the effect on glucose control of adding Welchol to an anti-diabetic medication regimen.

DETAILED DESCRIPTION:
To understand the effect of the addition of colesevelam HCl to oral agent therapy in individuals with type 2 diabetes on glycemic control by utilizing a novel technology, continuous glucose monitoring with ambulatory glucose profile analysis. To date there are no studies of this compound that have employed continuous glucose monitoring (CGM) with ambulatory glucose profile (AGP) analysis to obtain data that will detail the diurnal glucose patterns associated with this therapy. We plan to employ CGM at critical points throughout the study. AGP analysis will enable rapid assessment of the clinical status of the subject. Using statistically stable estimates of hourly values represented by five percentile curves AGP depicts glucose exposure, variability and stability. Previously, we have used AGP analysis to characterize glucose perturbations in individuals ranging from normal glucose tolerance to overt type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 and ≤75 years of age
* Clinical diagnosis of type 2 diabetes
* Currently treated with metformin, a sulfonylurea, or combination metformin/sulfonylurea; stable dose for ≥3 months
* HbA1c of 7.0-9.0% inclusive
* If taking lipid lowering medications, stable dose for >30 days

Exclusion Criteria:

* Taken oral or injected prednisone or cortisone medications in the previous 30 days. (Topical or inhaled steroids will not be considered excluded medications.)
* Current use of insulin or TZD's, or incretins
* LDL <70 mg/dL
* Serum triglycerides >500 mg/dL
* History of hypertriglyceridemia-induced pancreatitis
* History of gastrointestinal disorder such as dysphagia, swallowing disorder, intestinal motility disorder or prior bowel obstruction
* History or presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study
* Unable to follow the study protocol
* Unable to speak, read and write in English
* Pregnant, planning to become pregnant, breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger S. Mazze, PhD, Study Director — International Diabetes Center at Park Nicollet; Elinor S. Strock, APRN, BC, Principal Investigator — International Diabetes Center at Park Nicollet; Robert M. Cuddihy, MD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Bays HE, Goldberg RB, Truitt KE, Jones MR. Colesevelam hydrochloride therapy in patients with type 2 diabetes mellitus treated with metformin: glucose and lipid effects. Arch Intern Med. 2008 Oct 13;168(18):1975-83. doi: 10.1001/archinte.168.18.1975. PMID 18852398
- [Result] Mazze RS, Strock E, Wesley D, Borgman S, Morgan B, Bergenstal R, Cuddihy R. Characterizing glucose exposure for individuals with normal glucose tolerance using continuous glucose monitoring and ambulatory glucose profile analysis. Diabetes Technol Ther. 2008 Jun;10(3):149-59. doi: 10.1089/dia.2007.0293. PMID 18473688
- [Result] Goldberg RB, Fonseca VA, Truitt KE, Jones MR. Efficacy and safety of colesevelam in patients with type 2 diabetes mellitus and inadequate glycemic control receiving insulin-based therapy. Arch Intern Med. 2008 Jul 28;168(14):1531-40. doi: 10.1001/archinte.168.14.1531. PMID 18663165
- [Result] Mazze RS, Strock E, Borgman S, Wesley D, Stout P, Racchini J. Evaluating the accuracy, reliability, and clinical applicability of continuous glucose monitoring (CGM): Is CGM ready for real time? Diabetes Technol Ther. 2009 Jan;11(1):11-8. doi: 10.1089/dia.2008.0041. PMID 19132850
- [Result] Zieve FJ, Kalin MF, Schwartz SL, Jones MR, Bailey WL. Results of the glucose-lowering effect of WelChol study (GLOWS): a randomized, double-blind, placebo-controlled pilot study evaluating the effect of colesevelam hydrochloride on glycemic control in subjects with type 2 diabetes. Clin Ther. 2007 Jan;29(1):74-83. doi: 10.1016/j.clinthera.2007.01.003. PMID 17379048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Jan 2010 to Mar 2011. Medical Clinic Setting.
Groups:
- Welchol Then Placebo: 3.75 grams of colesevelam HCl (Welchol) taken for 12 weeks at evening meal, and then crossover to placebo taken at evening meal fro 12 weeks.
- Placebo Then Welchol: Placebo taken for 12 weeks at evening meal, and then crossover to 3.75 grams of colesevelam HCl taken at evening meal for 12 weeks.
Period: Overall Study
Arm/Group | Welchol Then Placebo | Placebo Then Welchol
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Welchol Then Placebo: 3.75 grams of colesevelam HCl taken at evening meal for 12 weeks, then crossover to placebo taken at evening meal for 12 weeks.
- Placebo Then Welchol: Placebo taken at evening meal for 12 weeks, then crossover to 3.75 grams of colesevelam HCl taken at evening meal for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Welchol Then Placebo | Placebo Then Welchol | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.4) | 59.5 (7.2) | 59.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
Total norm AUC average [Mean (Standard Deviation); unit: mg/(dL/hr) (normalized)] — Total norm HbA1c AUC was assessed by the CGM. The baseline CGM period started 14 days before randomization (visit 1) and concluded at randomization (visit 2). The data was then normalized.
  mg/(dL/hr) (normalized) | 162.2 (16.0) | 167.7 (25.9) | 164.8 (20.9)
Sleep norm Area under the curve average by group [Mean (Standard Deviation); unit: mg/(dL/hr) (normalized)] — Sleep norm HbA1c AUC was assessed by the CGM. The baseline CGM period started 14 days before randomization (visit 1) and concluded at randomization (visit 2). The data was then normalized.
  mg/(dL/hr) (normalized) | 157.1 (14.3) | 161.2 (23.4) | 159.1 (18.8)
Wake norm area under the curve average by group [Mean (Standard Deviation); unit: mg/(dL/hr) (normalized)] — Wake norm HbA1c AUC was assessed by the CGM. The baseline CGM period started 14 days before randomization (visit 1) and concluded at randomization (visit 2). The data was then normalized.
  mg/(dL/hr) (normalized) | 165.2 (17.8) | 170.0 (28.1) | 167.5 (22.8)
Hypoglycemia percentage of time <70 mg/dL average by group [Mean (Standard Deviation); unit: percentage of time <70 mg/dL] — Hypoglycemia percentage of time <70 mg/dL average by group was assessed by the CGM. The baseline CGM period started 14 days before randomization (visit 1) and concluded at randomization (visit 2).
  percentage of time <70 mg/dL | 0.4 (0.4) | 0.3 (0.6) | 0.4 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Total Norm AUC Average by Group (Normalized)
Description: Double Blinded CGM used for 2 week periods at the start of treatment 1, end of treatment 1, start of treatment 2, and end of treatment 2.
Time Frame: 2 week periods at the start of treatment 1, end of treatment 1, start of treatment 2, and end of treatment 2.
Measure: Mean (Standard Deviation); unit: mg/(dL/hr) normalized
Arm/Group | Welchol Then Placebo | Placebo Then Welchol
Number analyzed (Participants) | 11 | 10
mg/(dL/hr) normalized
  Start of Treatment 1 | 150.8 (10.8) | 175.9 (29.2)
  End of Treatment 1 | 149.9 (17.2) | 175.1 (27.4)
  Start of Treatment 2 | 163.2 (23.5) | 159.4 (23.9)
  End of Treatment 2 | 177.9 (33.2) | 159.4 (25.3)

2. Primary Outcome: Sleep Norm AUC Average by Group (Normalized)
Description: Overnight glucose captured by CGM.
Time Frame: 2 week periods at the start of treatment 1, end of treatment 1, start of treatment 2, and end of treatment 2.
Measure: Mean (Standard Deviation); unit: mg/(dL/hr) normalized
Groups:
- Welchol Then Placebo: 3.75 grams of colesevelam HCl (Welchol) at evening meal for 12 weeks, and then crossover to placebo at evening meal for 12 weeks.
  colesevelam HCl: 3.75 grams of colesevelam HCl (6 tablets)
  placebo
- Placebo Then Welchol: Placebo taken for 12 weeks at evening meal, and then crossover to 3.75 grams of colesevelam HCl taken at evening meal fro 12 weeks.
  colesevelam HCl: 3.75 grams of colesevelam HCl (6 tablets)
  placebo
Arm/Group | Welchol Then Placebo | Placebo Then Welchol
Number analyzed (Participants) | 11 | 10
mg/(dL/hr) normalized
  Start of Treatment 1 | 147.4 (16.6) | 161.9 (25.7)
  End of Treatment 1 | 148.0 (24.0) | 160.2 (27.9)
  Start of Treatment 2 | 158.8 (31.8) | 147.9 (24.4)
  End of Treatment 2 | 172.0 (32.5) | 143.6 (18.6)

3. Primary Outcome: Wake Norm AUC Average by Group (Normalized)
Description: Wake glucose captured by continuous glucose monitoring (CGM).
Time Frame: 2 week periods at the start of treatment 1, end of treatment 1, start of treatment 2, and end of treatment 2.
Measure: Mean (Standard Deviation); unit: mg/(dL/hr) (normalized)
Arm/Group | Welchol Then Placebo | Placebo Then Welchol
Number analyzed (Participants) | 11 | 10
mg/(dL/hr) (normalized)
  Start of Treatment 1 | 153.3 (11.7) | 180.9 (32.2)
  End of Treatment 1 | 151.2 (16.0) | 180.6 (29.6)
  Start of Treatment 2 | 165.2 (21.2) | 163.8 (25.6)
  End of Treatment 2 | 180.9 (34.2) | 165.2 (30.5)

4. Primary Outcome: Hypoglycemia Percentage of Time <70 mg/dL Average by Group
Description: Ambulatory glucose profile (AGP) reports were examined for the changes in the incidence of hypoglycemia (CGM<70 mg/dL)
Time Frame: 2 week periods at the start of treatment 1, end of treatment 1, start of treatment 2, and end of treatment 2.
Measure: Mean (Standard Deviation); unit: percentage of time <70 mg/dL
Arm/Group | Welchol Then Placebo | Placebo Then Welchol
Number analyzed (Participants) | 11 | 10
percentage of time <70 mg/dL
  Start of Treatment 1 | 1.2 (1.3) | 0.3 (0.6)
  End of Treatment 1 | 0.8 (1.1) | 0.4 (0.6)
  Start of Treatment 2 | 0.8 (1.2) | 0.7 (1.0)
  End of Treatment 2 | 0.6 (1.2) | 0.6 (1.1)

ADVERSE EVENTS:
Groups:
- Welchol: 3.75 grams of colesevelam HCl taken at evening meal
- Placebo: Placebo taken at evening meal
Arm/Group | Welchol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes